CLINICAL TRIAL: NCT05716906
Title: The Effects of Melatonin on Sleep Spindles in Children With Autism
Brief Title: Melatonin and Sleep Spindles in Autism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P002832
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Melatonin
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melatonin (Experimental): 5mg melatonin gummy 30 min before bedtime for 2 consecutive nights
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — 5mg gummy 30 min before bedtime for 2 consecutive nights

SUMMARY:
Sleep disturbances and sensory sensitivities are common disabling features of autism, but their underlying causes are not clear. We hypothesize that both of these difficulties reflect disrupted communication between a deep brain structure, the thalamus, and the brain's outer layer, the cortex. This communication is mediated by the thalamic reticular nucleus (TRN). Due to its small size and location deep in the brain, we cannot assess TRN function without invasive techniques. Fortunately, sleep spindles, a specific brain rhythm provide a noninvasive read-out of TRN function. In Aim 1 we will examine whether reduced sleep spindles are related to worse sleep quality, impaired selective attention during wake, and sensory sensitivities in children with autism. In Aim 2, we will determine whether melatonin, which is commonly used to improve sleep, also increases sleep spindles in autism. If successful, this study will introduce TRN as a target for treatment of sleep disruption and guide larger home-based sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with ASD
* 12-18 years of age
* English speaking
* Able to understand and respond to questionnaires in English

Exclusion Criteria:

* Pregnant or breastfeeding
* Substance abuse or dependence within the past six months (nicotine abuse or dependence is not exclusionary)
* Chronic medical conditions that affect sleep
* Any unstable chronic medical condition such as asthma, diabetes, cystic fibrosis, or cardiac disease
* History of head injury resulting in prolonged loss of consciousness or other neurological sequelae
* IQ <70
* Other neurological disorder, including seizure disorder
* Diagnosed sleep disorder
* Known genetic causes of ASD
* Currently taking melatonin or those who have had an adverse reaction to melatonin in the past

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sleep spindle density | Five nights of sleep over two weeks
  Changes in sleep spindle density (#/min) during non-Rapid Eye Movement (NREM) sleep between baseline and melatonin nights as measured by portable EEG device.

SECONDARY OUTCOMES:
Change in sleep quality | Five nights of sleep over two weeks
  Change in sleep quality between baseline and melatonin nights

CONTACTS AND LOCATIONS:
Overall Officials: Dara Manoach, PhD, Principal Investigator — Professor
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will disseminate results through presentations at public lectures, scientific institutions and meetings, and/or publications in major journals. Specifically, quality-controlled data used in publications will be deidentified and made available to requesting scientists, after publication of the results. Workflows will be documented and will allow any external groups to reproduce results from the raw data.
Time Frame: Data will be available following the publication of the results.